CLINICAL TRIAL: NCT05476120
Title: The Effect of the Use of BATHE Interview Technique on Treatment Compliance in Hypertension Patients in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Vildan Mevsim, Prof.Dr., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Duygu ATALI
Record Dates: First submitted 2021-11-14; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Intervention Model Description: single-blind, parallel-group, randomized-controlled intervention study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BATHE (Experimental): In each interview, the intervention group was intervened by the physician to increase compliance with the treatment using the BATHE technique, and brief information was given emphasizing the importance of drug compliance and lifestyle changes routinely applied by the Family Medicine Department in hypertension patients. The patients in the intervention group were interviewed face-to-face at the 0th and 6th months, and online at the 3rd month.
  Interventions: Behavioral: BATHE
- Control (No Intervention): In the control group, brief information was given at each interview, emphasizing the importance of drug compliance and lifestyle changes routinely applied by the Department of Family Medicine in hypertension patients. No intervention was made. The patients in the control group were interviewed face-to-face at 0 and 6 months, and online at 3 months.

INTERVENTIONS:
Behavioral: BATHE — The BATHE interview technique was applied 3 times, once every 3 months, for 6 months.
  Arms: BATHE

SUMMARY:
The research is planned to evaluate the treatment compliance after the BATHE interview technique in hypertension patients.

DETAILED DESCRIPTION:
In order to be evaluated for suitability for the study, patients aged 18-80 who have been diagnosed with hypertension for at least 6 months (n= 220) were interviewed and 86 hypertension patients who met the inclusion criteria and volunteered for the study were included in the study. Participants whose eligibility was determined as a result of the evaluation in terms of inclusion and exclusion criteria were asked about their volunteerism in the intervention study, their written consent was obtained from those who volunteered, and those who volunteered were randomized.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient of hypertension
* Be over 18 years old
* Be less than 80 years old
* To have been diagnosed for at least 6 months
* Volunteering
* To be able to use any of the online video calling channels

Exclusion Criteria:

* Communication problem
* Presence of psychiatric illness and/or use of psychiatric medication
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The Scale for Evaluating the Success of Treatment Adherence and Lifestyle Change in Hypertensive Individuals | Baseline and sixth month
  The scale consists of 18 questions. The questions were structured in a positive and negative way and the answers were expressed as a five-point likert. The contents of the questions were prepared to enlighten the subjects of medical treatment and clinical controls, communication with the physician, active lifestyle and physical activity, weight control, healthy nutrition and salt consumption, and disease awareness. After reverse scoring, if all items are given 5 points, the highest total score that can be obtained from the scale is 90. When all items are given 1 point, the lowest score that can be obtained from the scale is 18. The scale cutoff point is 68. A score of less than 68 indicates low adherence to treatment, and a score of 68 and above indicates high adherence to treatment. An increase in the score on the scale indicates an increase in treatment compliance.
Turkish Modified Morisky Scale | Baseline and sixth month
  The scale consists of 6 questions. The questions were answered as Yes/No and in the evaluation; in questions 2 and 5 yes 1 point, no 0 points; In other questions, yes is 0 points, no is 1 point. If the total score obtained by the patient in questions 1, 2 and 6 is 0 or 1, it indicates low motivation level, and >1 indicates high motivation level. If the total score from questions 3, 4 and 5 is 0 or 1, it indicates low level of knowledge, and >1 indicates high level of knowledge.

SECONDARY OUTCOMES:
Waist circumference | Baseline and sixth month
  At the beginning and at the 6th month, the waist circumference of the participants was measured by the researcher under appropriate conditions and in both interviews.
BMI | Baseline and sixth month
  At the beginning and at the 6th month, BMI of the participants was measured by the researcher under appropriate conditions and in both interviews.
Blood pressure | Baseline and sixth month
  In both interviews, both systolic and diastolic blood pressures of the participants were measured by the researcher under appropriate conditions and at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Vildan MEVSİM, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No